CLINICAL TRIAL: NCT07075354
Title: Clinical and Radiographic Outcomes of Root Canal Obturation With Hydraulic Condensation and Bioceramic Biomaterial: A 12-Month Prospective Study on Periapical Healing
Brief Title: Healing Outcomes Following Hydraulic Condensation With a Bioactive Bioceramic Sealer in Root Canal Treatment
Acronym: HEAL-BR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Plovdiv Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MU-Endo-HCBR2021-01
Record Dates: First submitted 2025-07-01; First posted 2025-07-20 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Irreversible Pulpitis; Apical Periodontitis
Keywords: bioceramic sealer; BioRoot RCS; hydraulic condensation; periapical healing; PAI
MeSH Terms: conditions — Periapical Periodontitis

STUDY DESIGN:
Intervention Model Description: This is a single-group assignment interventional study assessing the healing outcomes of root canal treatment using hydraulic condensation with the bioceramic sealer BioRoot RCS. All participants receive the same standardized treatment protocol and are followed prospectively for 12 months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hydraulic Condensation with BioRoot RCS (Experimental): This arm involves root canal treatment using the hydraulic condensation technique combined with BioRoot RCS, a bioceramic calcium silicate-based sealer. The procedure includes standardized irrigation with sonic activation, drying using a single calibrated paper point without alcohol, and single-visit obturation. BioRoot RCS sets hydraulically in the presence of moisture, promotes hard tissue formation, and provides a durable seal to support periapical healing.
  Interventions: Procedure: Hydraulic Condensation Root Canal Obturation with BioRoot RCS

INTERVENTIONS:
Procedure: Hydraulic Condensation Root Canal Obturation with BioRoot RCS — Root canal obturation using the hydraulic condensation technique combined with BioRoot RCS, a bioceramic calcium silicate-based sealer. Treatment includes standardized irrigation with sonic activation and drying using a single calibrated paper point without alcohol. The sealer sets hydraulically in the presence of moisture, promotes hard tissue formation, and provides a durable, bioactive seal supporting periapical healing.
  Other Names: BioRoot RCS bioceramic sealer; Calcium silicate-based root canal sealer

SUMMARY:
This prospective clinical study aimed to evaluate the healing outcomes after root canal treatment using a bioceramic sealer called BioRoot RCS in combination with a technique known as hydraulic condensation. Root canal treatment is a common procedure used to remove infection and preserve teeth. Bioceramic materials have recently gained attention due to their ability to support natural healing, form a strong seal in the root canal, and stimulate tissue regeneration.

A total of 66 permanent teeth from patients diagnosed with either irreversible pulpitis or apical periodontitis were treated and followed over a 12-month period. All treatments were completed in a single visit and followed a standardized protocol using sonic irrigation and a calibrated drying method. The sealer used-BioRoot RCS-is a bioactive, calcium silicate-based material that hardens in the presence of moisture and promotes healing.

Patients were monitored clinically and radiographically using the Periapical Index (PAI), which is a scale that measures the status of periapical tissue (area around the root tip). Healing was considered successful if the treated teeth remained symptom-free and showed favorable radiographic changes over time.

DETAILED DESCRIPTION:
This prospective single-arm clinical study was designed to evaluate the healing outcomes following root canal treatment performed using a calcium silicate-based bioceramic sealer (BioRoot™ RCS) in conjunction with the hydraulic condensation obturation technique. The protocol emphasized clinical standardization, with all treatments completed in a single visit by experienced endodontists under magnification.

Following local anesthesia and rubber dam isolation, root canals were prepared using rotary nickel-titanium instrumentation to a standardized apical size (generally ISO 35-45 depending on canal anatomy), and irrigation was performed with 5.25% sodium hypochlorite (NaOCl) activated with a sonic device (EndoActivator, Dentsply Sirona). A final rinse protocol included 17% EDTA and saline, followed by calibrated drying with a single paper point to ensure optimal moisture conditions for the setting of the bioceramic sealer.

BioRoot RCS was mixed according to the manufacturer's instructions and delivered into the canals using a dedicated syringe tip. A single-cone gutta-percha point matching the apical preparation size was inserted with slight apical pressure to displace excess sealer, completing the hydraulic condensation process. No thermoplasticized techniques or heat sources were used to preserve the bioactive potential of the sealer.

Postoperative radiographs were taken immediately and at recall intervals of 6 and 12 months. Clinical and radiographic evaluations were conducted using the Periapical Index (PAI), with scoring by two calibrated examiners blinded to the clinical data. Inter-examiner agreement was assessed using Cohen's kappa.

The primary endpoint was periapical healing, operationally defined as a reduction in PAI score and the absence of symptoms. Comparative analysis was also performed between teeth with and without baseline periapical pathology to assess differential healing responses.

ELIGIBILITY:
The inclusion criteria encompassed:

permanent teeth patients aged over 18 years both biological genders good general health, teeth diagnosed with irreversible pulpitis or apical periodontitis

Exclusion criteria included:

teeth with previous root canal treatment, teeth with open apices (immature teeth), teeth with extensive resorption, teeth with severe periodontal disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2021-01-20 (Actual); Primary Completion 2022-01-20 (Actual); Study Completion 2022-01-20 (Actual)

PRIMARY OUTCOMES:
Periapical Healing Assessed by Periapical Index (PAI) Score | Baseline, 6 months, and 12 months post-treatment
  Radiographic assessment of periapical healing using the Periapical Index (PAI) scoring system on standardized periapical radiographs. Successful healing is defined as a reduction in PAI score indicating resolution or significant improvement of apical periodontitis.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Plovdiv, Faculty of Dental Medicine, Department of Operative Dentistry and Endodontics, Plovdiv, Plovdiv, Bulgaria

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) will be made available to qualified researchers upon reasonable request. Data sharing will follow institutional and ethical guidelines, ensuring participant confidentiality. Access will be granted after publication of the main study results and completion of any necessary data use agreements.
Supporting Information: Study Protocol, ICF
Time Frame: The individual participant data (IPD) and supporting documentation will be available starting 6 months after publication of the main study results and will remain accessible for a period of 5 years.
Access Criteria: Qualified researchers who submit a reasonable research proposal will be granted access to de-identified IPD and supporting materials. Requests will be reviewed by the study investigators and institutional review board to ensure ethical use and protection of participant privacy. Data will be shared via a secure data transfer platform following signing of a data use agreement.